CLINICAL TRIAL: NCT06905678
Title: The Financial and Emotional Impact of Cleft Palate on Children and Their Caregivers: a Mixed-method Study
Brief Title: The Financial and Emotional Impact of Cleft Palate
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0282
Record Dates: First submitted 2024-11-28; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cleft Lip and Cleft Palate
Keywords: Cleft lip and palate; Emotional burden; Financial burden; Questionnaires; Perceptions; Interviews
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Financial Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Children/young adults with cleft lip and/or palate: This group are children and young adults with a cleft lip and/or a cleft palate. They are 5, 12 or 22 years old.
  Interventions: Other: Questionnaires; Other: Semi-structured interviews
- Children/young adults without a cleft: This group consists of healthy children and young adults. They will be age and gender matched to the group of children/young adults with a cleft.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The participants will fin in questionnaires about the financial and emotional burden they experience.
Other: Semi-structured interviews — After the participants have filled in the questionnaires they will get the chance to participate in an interview to talk about their perceptions and experiences.
  Groups: Children/young adults with cleft lip and/or palate

SUMMARY:
Cleft lip and/or palate (CL±P) is the most prevalent congenital craniofacial defect with a significant social impact, affecting speech, hearing, feeding, oral behavior, dentition and satisfaction with appearance. These consequences have a long-term and negative impact on social integration and well-being. WHO highlights the significant financial costs, including morbidity, healthcare costs, emotional distress and social exclusion to patients, their families and society. The purpose of this study is to investigate the financial and emotional impact of CL±P based on the perceptions of children with CL±P and their parents/guardians followed by the interdisciplinary craniofacial teams of the University Hospitals of Leuven or Ghent. Participation in this study consists of completing questionnaires related to financial, social and well-being aspects using the CLEFT-Q, Parental Stress Scale and a financial impact questionnaire. The parents/guardians of the children aged 5 years always complete all questionnaires. The parents/guardians of the 12- and 18-year-old children complete the Parental Stress Scale and a financial impact questionnaire. The children aged 18 complete the CLEFT-Q themselves. Questionnaires can be delivered online or on paper. The outcomes on the health-related QoL of children with cleft and the PSS are compared with the outcomes of 'healthy' children and their parents/guardians to ensure that the emotional impact is attributable to the cleft. In addition, children and their parents/guardians can participate in a semi-structured interview. During the interview appointment, the questionnaires can be completed on paper. Potential participants will be told that the interview will be recorded and that all findings will be kept confidential. The actual interviews will take place at a location and time that is most convenient for the participants. Participants do not need to come to UZ Gent or UZ Leuven for this. Each interview will be recorded with a Roland R-05 high quality audio recorder. After conducting the interviews, all participants will be asked to complete a questionnaire regarding their demographic data. In addition, data regarding the type of cleft, diagnoses, observation sheets and consultation letters will be collected from the medical records of the children with CL±P. We also aim to investigate whether variations in these effects are observable based on the specific type of cleft. All participants will go through the same protocol regardless of recruitment through UZ Gent or UZ Leuven.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a cleft (lip and) palate
* Age of 5, 12 or 18 years

Exclusion Criteria:

- No specific exclusion criteria

Ages: 4 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population are children/young adults with a cleft (lip and) palate and their parents/caregivers. To verify some results a control group is included consisting of healthy children/young adults and their parents/caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Financial burden of a cleft | 2 months
  The parents of children with a cleft will fill in a questionnaire regarding the costs of having a child with a cleft. Using this information and de electronic patient record the investigators can calculate the estimated cost of having a child with a cleft.
Emotional burden of a cleft | 2 months
  Using questionnaires the emotional burden of a cleft will be examined. The parents of the children with a cleft will fill in the Parental Stress Scale (18 items that evaluate parents' feelings about their parental role, with both positive and negative aspects of parenting), and the children with a cleft will fill in the CLEFT-Q (a comprehensive Patient-Reported Outcome Measure (PROM) evaluating QoL, facial function and assessment of appearance).

SECONDARY OUTCOMES:
Differences in impact based on the type of cleft | Through study completion, an average of 1 year
  The investigators want to examine if the results on the questionnaire will be different based on the type of cleft. Participants filled in the questionnaires on which type of cleft they have. The results are then reviewed and compared to see if the results obtained depend on the type of cleft.
Does the impact decrease as the child gets older | Through study completion, an average of 1 year
  The investigators want to examine if the financial and emotional burden decreases as the child gets older by comparing the financial and emotional impact of the different ages of children/young adults included. For this purpose, the results on the questionnaires of the 3 age groups will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No